CLINICAL TRIAL: NCT02908854
Title: Using Spices and Herbs to Increase Vegetable Intake Among Urban High School Students in the National School Lunch Program
Brief Title: Using Spices and Herbs to Increase Vegetable Intake Among Urban High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Chris D'Adamo, Director of Research Center for Integrative Medicine, University of Maryland, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00066121
Record Dates: First submitted 2016-09-07; First posted 2016-09-21 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Poor Nutrition
Keywords: Spices; Herbs; Vegetables; National School Lunch Program; High school
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- School Lunch Participants (Experimental): School lunch participants will be given vegetables with and without additional spices and herbs to determine if intake will increase with the addition of spices and herbs.
  Interventions: Other: Adding spices and herbs to school lunch vegetables

INTERVENTIONS:
Other: Adding spices and herbs to school lunch vegetables — Direct measurement of school lunch vegetable intake among students both before and after spices and herbs are added.

SUMMARY:
A two-phase, school-based intervention will be conducted at a high school in Baltimore to evaluate whether the addition of spices and herbs to vegetable dishes in the National School Lunch Program (NSLP) can increase vegetable intake among students in an urban and predominantly African-American high school.

DETAILED DESCRIPTION:
The proposed research will be conducted at Cristo Rey Jesuit High School in Baltimore, Maryland. In this two-phase intervention, the research team will work in Phase I with stakeholders throughout the high school community to identify the barriers to vegetable intake in the NSLP in this student population and to determine how spices and herbs might help overcome these barriers. The stakeholders with whom we will collaborate will include students, school administration, and cafeteria staff.

Phase II will focus on the direct measurement of vegetable intake among students both before and after spices and herbs are added to the vegetables in the NSLP. The spiced vegetable recipes that received the most favorable student rankings in the taste tests of Phase I will be offered.

The vegetable recipes flavored with spices and herbs will meet all NSLP requirements for fat, sugar, total calories, and all other guidelines.

Student vegetable intake will be assessed through two outcomes: 1.) plate waste, and 2.) production waste.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled student at Cristo Rey High School
* Able to read and write English (exclusive to Phase 1 participants)

Exclusion Criteria:

* Does not eat lunch in the Cristo Rey High School cafeteria
* Not willing to complete questionnaires (exclusive to Phase 1 participants)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Vegetable plate waste | The overall time frame for the outcome measure assessment is up to 8 months. This will occur during the 2016-2017 school year.
  Student vegetable intake will be assessed through plate waste (weighed).

SECONDARY OUTCOMES:
Cafeteria production waste as measured by calculating the difference between total prepared vegetable weight and discarded vegetable weight. | The overall time frame for the outcome measure assessment is up to 8 months. This will occur during the 2016-2017 school year.
  This outcome involves quantifying both the amount of vegetables that were prepared and served and the amount of vegetables that were thrown away by cafeteria staff after lunch.
Attitudes towards eating vegetables | The outcome measure is being assessed up to 12 months. Spring 2016 through Spring 2017.
  Participants will complete a baseline questionnaire in the Spring of 2016 followed by a follow-up questionnaire at the end of the 2016-2017 school year. Changes in attitudes towards eating vegetables will be assessed before and after the addition of spices and herbs to the school lunch vegetables.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D'Adamo, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Center for Integrative Medicine University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gase LN, McCarthy WJ, Robles B, Kuo T. Student receptivity to new school meal offerings: assessing fruit and vegetable waste among middle school students in the Los Angeles Unified School District. Prev Med. 2014 Oct;67 Suppl 1(0 1):S28-33. doi: 10.1016/j.ypmed.2014.04.013. Epub 2014 Apr 16. PMID 24747044
- [Background] Byker CJ, Farris AR, Marcenelle M, Davis GC, Serrano EL. Food waste in a school nutrition program after implementation of new lunch program guidelines. J Nutr Educ Behav. 2014 Sep-Oct;46(5):406-11. doi: 10.1016/j.jneb.2014.03.009. Epub 2014 May 22. PMID 24857599
- [Background] Just DR, Wansink B, Hanks AS. Chefs move to schools. A pilot examination of how chef-created dishes can increase school lunch participation and fruit and vegetable intake. Appetite. 2014 Dec;83:242-247. doi: 10.1016/j.appet.2014.08.033. Epub 2014 Aug 27. PMID 25173063
- [Background] Hanks AS, Wansink B, Just DR. Reliability and accuracy of real-time visualization techniques for measuring school cafeteria tray waste: validating the quarter-waste method. J Acad Nutr Diet. 2014 Mar;114(3):470-474. doi: 10.1016/j.jand.2013.08.013. Epub 2013 Oct 14. PMID 24135053
- [Background] D'Adamo CR, McArdle PF, Balick L, Peisach E, Ferguson T, Diehl A, Bustad K, Bowden B, Pierce BA, Berman BM. Spice MyPlate: Nutrition Education Focusing Upon Spices and Herbs Improved Diet Quality and Attitudes Among Urban High School Students. Am J Health Promot. 2016 May;30(5):346-56. doi: 10.1177/0890117116646333. PMID 27404643